CLINICAL TRIAL: NCT06729216
Title: Species Identification and Antifungal Susceptibility Testing of Dermatophytes Isolated From Patients Attending Dermatology Outpatient Clinic at Kasr Alainy Hospitals
Brief Title: Fungal Resistance in Dermatophyte Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, University doctor, Cairo University
Other Study IDs: Cutaneous Fungal resistance
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Dermatophyte Infection
MeSH Terms: conditions — Dermatomycoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antifungal susceptibility testing (AFST)
  Interventions: Diagnostic Test: Antifungal susceptibility testing (AFST)

INTERVENTIONS:
Diagnostic Test: Antifungal susceptibility testing (AFST) — testing the fungal susceptibility to different drugs

SUMMARY:
The aim of the study is to compare the efficiency of broth microdilution versus disk diffusion method for antifungal drug susceptibility testing of the most used drugs in dermatophytosis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed clinically with dermatophytosis, any age group and any sex

Exclusion Criteria:

* Patients under either Local or systemic antifungal treatment

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with dermatophytic skin infection
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Precent susceptibility to each drug | 3 months
  Measure the area of inhibition zone of the drugs to the fungus on the culture